CLINICAL TRIAL: NCT00252031
Title: Dialectical Behavioral Therapy for Patients With Borderline Personality Disorder
Brief Title: DBT in Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3277-02-0002
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2005-11-21 (Estimated); Status verified 2005-11

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; BPD; Dialectical Behavior Therapy; DBT
MeSH Terms: conditions — Borderline Personality Disorder

INTERVENTIONS:
Behavioral: Dialectical Behavioral Therapy

SUMMARY:
Subjects will receive a 6-month course of DBT, consisting of one 90-minute group and one 60-minute individual session per week as well as telephone availability of the individual therapist.

ELIGIBILITY:
Inclusion Criteria: Is a male or female between 18 and 60 who meets criteria for Borderline Personality Disorder and has had at least 2 prior instances of suicidal or parasuicidal behavior. Either is off psychotropic drugs or is on a stable medication regimen. (During the study, psychotropic medications will be prescribed by a psychiatrist in the Mood and Personality Disorders Group.)

Exclusion Criteria: Meets criteria for Schizophrenia, Bipolar Disorder, Mental Retardation or current or recent Substance Dependence. Subjects also should not currently be in individual psychotherapy. (Case management and work therapy programs are allowed.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Measures of parasuicidal behavior, suicidal ideation, mood and emotion, dissociation and health care utilization at baseline, 3 months, 6 months and 9 months

SECONDARY OUTCOMES:
Measures of cognitive processing at baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Goodman, MD, Principal Investigator — Bronx VA Medical Center/Mount Sinai School of Medicine
Locations (1):
- Bronx VA Medical Center, The Bronx, New York, United States